CLINICAL TRIAL: NCT00305409
Title: Synbiotic Treatment in Crohn's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CZB/4/335; RND ID: 2004GA07; LREC Ref: 05/51401/111
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's; TNF-alpha; Synbiotic; Probiotic
MeSH Terms: conditions — Crohn Disease | interventions — Synbiotics

INTERVENTIONS:
Drug: Synbiotic (Synergy I / B.longum)

SUMMARY:
The purpose of this study is to determine whether administration of a synbiotic, comprised on inulin and a bifidobacterial probiotic will colonise the gut wall and down-regulate TNF-alpha and other pro-inflammatory cytokines in the mucosa of Crohn's patients with active disease to reduce mucosal inflammation and induce remission.

DETAILED DESCRIPTION:
Crohn's disease is one of the two main forms of idiopathic inflammatory bowel disease. The Th1-mediated inflammatory response in Crohn's disease is characterised by increased IL-18 and INF-gamma and especially TNF-alpha, which are formed by lamina propria mononuclear cells. The aim of this investigation is to determine whether a synbiotic comprised of inulin and a bifidobacterial probiotic, that we have previously shown to down-regulate TNF-alpha and other proinflammatory cytokines in the gut mucosa in ulcerative colitis patients with active disease, can colonise the bowel wall, reduce mucosal inflammation and induce remission in Crohn's disease patients with active disease, in a randomised controlled trial. Crohn's disease is associated with high mortality and incurs significant social, commercial and NHS costs. Many patients are refractile to standard treatments, which often have undesirable side effects. An inexpensive, effective and non-toxic treatment based on the synbiotic concept would contribute greatly to relieving the clinical and financial burdens of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease of large bowel (+/- small bowel disease)
* 18-79 years old
* stable doses of medications
* CDAI >150, <450

Exclusion Criteria:

* short gut syndrome
* pregnancy
* lactation
* antibiotic therapy in last 3 months
* probiotic therapy in last 1 month
* <18, >79 years old
* CDAI <150 or >450
* indeterminate colitis, ulcerative colitis
* alterations to medications in last 3 months

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Reduction in mucosal TNF-alpha

SECONDARY OUTCOMES:
Number of patients in remission as assessed by CDAI.
Significant differences in mucosal regeneration between pre-synbiotic and post-synbiotic therapy groups and pre-control and post-control therapy groups.
Differences in TNF-alpha, IL-18 and INF-gamma between the post-synbiotic and post-control groups.

CONTACTS AND LOCATIONS:
Overall Officials: George MacFarlane, BSc PhD, Principal Investigator — University of Dundee
Locations (2):
- United Kingdom (2):
  - Dundee University, Dept of Pathology and Neuroscience, Dundee, Angus
  - Ninewells Hospital and Medical School, Dundee, Tayside

REFERENCES:
- [Background] Furrie E, Macfarlane S, Kennedy A, Cummings JH, Walsh SV, O'neil DA, Macfarlane GT. Synbiotic therapy (Bifidobacterium longum/Synergy 1) initiates resolution of inflammation in patients with active ulcerative colitis: a randomised controlled pilot trial. Gut. 2005 Feb;54(2):242-9. doi: 10.1136/gut.2004.044834. PMID 15647189
- [Background] Fite A, Macfarlane GT, Cummings JH, Hopkins MJ, Kong SC, Furrie E, Macfarlane S. Identification and quantitation of mucosal and faecal desulfovibrios using real time polymerase chain reaction. Gut. 2004 Apr;53(4):523-9. doi: 10.1136/gut.2003.031245. PMID 15016746
- [Background] Bartosch S, Woodmansey EJ, Paterson JC, McMurdo ME, Macfarlane GT. Microbiological effects of consuming a synbiotic containing Bifidobacterium bifidum, Bifidobacterium lactis, and oligofructose in elderly persons, determined by real-time polymerase chain reaction and counting of viable bacteria. Clin Infect Dis. 2005 Jan 1;40(1):28-37. doi: 10.1086/426027. Epub 2004 Dec 6. PMID 15614689
- [Background] Macfarlane GT, Cummings JH. Probiotics and prebiotics: can regulating the activities of intestinal bacteria benefit health? BMJ. 1999 Apr 10;318(7189):999-1003. doi: 10.1136/bmj.318.7189.999. No abstract available. PMID 10195977
- [Background] Bassi A, Dodd S, Williamson P, Bodger K. Cost of illness of inflammatory bowel disease in the UK: a single centre retrospective study. Gut. 2004 Oct;53(10):1471-8. doi: 10.1136/gut.2004.041616. PMID 15361497
- [Background] Stange EF, Travis SP, Vermeire S, Beglinger C, Kupcinkas L, Geboes K, Barakauskiene A, Villanacci V, Von Herbay A, Warren BF, Gasche C, Tilg H, Schreiber SW, Scholmerich J, Reinisch W; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: definitions and diagnosis. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i1-15. doi: 10.1136/gut.2005.081950a. No abstract available. PMID 16481628
- [Background] Furrie E, Macfarlane S, Cummings JH, Macfarlane GT. Systemic antibodies towards mucosal bacteria in ulcerative colitis and Crohn's disease differentially activate the innate immune response. Gut. 2004 Jan;53(1):91-8. doi: 10.1136/gut.53.1.91. PMID 14684582
- [Background] Caprilli R, Gassull MA, Escher JC, Moser G, Munkholm P, Forbes A, Hommes DW, Lochs H, Angelucci E, Cocco A, Vucelic B, Hildebrand H, Kolacek S, Riis L, Lukas M, de Franchis R, Hamilton M, Jantschek G, Michetti P, O'Morain C, Anwar MM, Freitas JL, Mouzas IA, Baert F, Mitchell R, Hawkey CJ; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: special situations. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i36-58. doi: 10.1136/gut.2005.081950c. PMID 16481630
- [Background] Travis SP, Stange EF, Lemann M, Oresland T, Chowers Y, Forbes A, D'Haens G, Kitis G, Cortot A, Prantera C, Marteau P, Colombel JF, Gionchetti P, Bouhnik Y, Tiret E, Kroesen J, Starlinger M, Mortensen NJ; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: current management. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i16-35. doi: 10.1136/gut.2005.081950b. PMID 16481629